CLINICAL TRIAL: NCT01808118
Title: A Multicenter, Randomized, Double-Blind, Study Comparing the Efficacy and Safety of Continuing Versus Withdrawing Adalimumab Therapy in Maintaining Remission in Subjects With Non-Radiographic Axial Spondyloarthritis
Brief Title: Continuing Versus Withdrawing Adalimumab in Maintaining Remission in Non-Radiographic Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-375; 2012-000646-35 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Axial Spondyloarthritis
Keywords: Spondylitis; Spondylarthropathy; Ankylosing Spondyloarthritis; Spondyloarthritis; Spinal Diseases; Musculoskeletal Diseases; Arthritis; Joint Diseases; Adalimumab; Antirheumatic Agents; Anti-Inflammatory Agents
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis; Spondylarthropathies; Spondylitis, Ankylosing; Spondylarthritis; Spinal Diseases; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-Blind Adalimumab (Experimental): 40 mg every other week (eow), Weeks 28-68. Blinded adalimumab was discontinued in participants who met the criteria for flare.
  Interventions: Biological: adalimumab
- Open-label (OL) Adalimumab (Experimental): 40 mg every other week (eow), Weeks 0-28. If participants flared during the double-blind period, they had an opportunity to receive at least 12 weeks of open-label adalimumab 40 mg eow.
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator): Placebo every other week (eow), Weeks 28-68. Placebo was discontinued in participants who met the criteria for flare.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: adalimumab — 40 mg every other week
  Other Names: Humira; ABT-D2E7
  Arms: Double-Blind Adalimumab; Open-label (OL) Adalimumab
Biological: Placebo — every other week
  Arms: Placebo

SUMMARY:
The objective of this multicenter, randomized, double-blind study was to evaluate the efficacy and safety of continuing versus withdrawing therapy with adalimumab 40 mg given every other week SC in maintaining remission in subjects with moderate to severe non-radiographic axial spondyloarthritis.

DETAILED DESCRIPTION:
The study duration included a 42-day Screening Period, a 28-week open-label 40 mg adalimumab every other week (eow) treatment period (Period 1), a 40-week double-blind placebo controlled eow treatment period (Period 2) with an opportunity to receive at least 12 weeks of rescue therapy with open-label adalimumab (participants that flared at Weeks 60, 64 or 68 were allowed 12 weeks of rescue therapy and final visits were at Weeks 72, 76 or 80 respectively), plus a 70-day follow-up phone call. Participants in sustained Ankylosing Spondylitis Disease Activity Score (ASDAS) inactive disease were randomized at Week 28 at a 1:1 ratio to receive either blinded adalimumab 40 mg eow or matching placebo. The length of exposure to adalimumab depended on remission or flare status and ranged from 20 (first time Ankylosing Spondylitis Disease Activity Score [ASDAS] remission was calculated) to 80 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with inadequate response to ≥2 nonsteroidal anti-inflammatory drugs (NSAIDs)
* Participants with non-radiographic axial spondyloarthritis fulfilling the Assessment of Spondyloarthritis International Society (ASAS) axial SpA classification criteria, but not fulfilling the radiologic criterion of the modified New York criteria for ankylosing spondylitis
* Participants must have baseline disease activity as defined by having an Ankylosing Spondylitis Disease Activity Score (ASDAS) ≥ 2.100, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4 and Patient's Assessment of Total Back Pain score ≥ 4 based on a Numeric Rating Scale (NRS) at both the screening and baseline visits
* Participants with evidence of active inflammation in the sacroiliac (SI) joints or spine on MRI, or elevated high sensitivity C-reactive protein (hs-CRP) at screening
* Negative tuberculosis (TB) screening assessment
* Ability to administer subcutaneous injections or have a qualified person available to administer injections
* If female, either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy) or of childbearing potential and practicing an approved method of birth control throughout the study and for 150 days after last dose of study drug.
* Participant judged to be in good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, chest X-ray, and a 12-lead electrocardiogram performed at screening

Exclusion Criteria:

* Prior anti-Tumor Necrosis Factor (TNF) therapy; biologic therapy with a potential therapeutic impact on SpA or treated with an investigational drug of chemical or biologic nature within 30 days or 5 half-lives prior to the baseline visit.
* Fulfillment of the radiologic criterion of the modified New York criteria for Ankylosing Spondylitis at or prior to the screening visit
* Recent infection requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the baseline visit or oral anti-infectives within 14 days prior to the baseline visit
* Significant medical events or conditions that may put participants at risk for participation
* Female participants who are pregnant or breast-feeding or considering becoming pregnant during the study
* Known hypersensitivity to adalimumab or its excipients as stated in the label

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landewe R, Sieper J, Mease P, Inman RD, Lambert RG, Deodhar A, Marzo-Ortega H, Magrey M, Kiltz U, Wang X, Li M, Zhong S, Mostafa NM, Lertratanakul A, Pangan AL, Anderson JK. Efficacy and safety of continuing versus withdrawing adalimumab therapy in maintaining remission in patients with non-radiographic axial spondyloarthritis (ABILITY-3): a multicentre, randomised, double-blind study. Lancet. 2018 Jul 14;392(10142):134-144. doi: 10.1016/S0140-6736(18)31362-X. Epub 2018 Jun 29. PMID 29961640
- See also: Humira Prescribing Information — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 42-day screening period.The Full Analysis Set (FAS) included all participants who enrolled in the open-label period (Period 1) and received at least 1 dose of adalimumab. The All Randomized Set included all Period 2 participants who were randomized to receive either placebo or 40 mg adalimumab every other week.
Groups:
- Open-label (OL) Adalimumab (Period 1): 40 mg every other week (eow), Weeks 0-28.
- Placebo (Period 2): Placebo every other week (eow), Weeks 28-68. Placebo was discontinued in participants who met the criteria for flare.
- Double-blind Adalimumab (Period 2): Adalimumab 40 mg every other week (eow), Weeks 28-68. Blinded adalimumab was discontinued in participants who met the criteria for flare.
Period: Period 1
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Started | 673 | 0 | 0
Completed | 305 | 0 | 0
Not Completed | 368 | 0 | 0
Not completed — Adverse Event | 15 | 0 | 0
Not completed — Withdrew consent | 24 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0
Not completed — Did not meet criteria for remission | 303 | 0 | 0
Not completed — Enrolled in error | 7 | 0 | 0
Not completed — Did not meet inclusion criteria | 3 | 0 | 0
Not completed — Non-conformance with inclusion criteria | 3 | 0 | 0
Not completed — Investigator decision: site closure | 2 | 0 | 0
Not completed — Non-compliance per sponsor | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Period 2
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Started | 0 | 153 | 152
Completed | 0 | 140 | 144
Not Completed | 0 | 13 | 8
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Withdrew consent | 0 | 7 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Investigator no longer conducting trials | 0 | 1 | 0
Not completed — Switched to other therapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who enrolled in the open-label period (Period 1) and received at least 1 dose of adalimumab.
Arm/Group | Open-label (OL) Adalimumab (Period 1)
Number analyzed (Participants) | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343
  Male | 330
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 651
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Did Not Experience a Flare During Period 2 by Week 68
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of high-sensitivity C-reactive protein (mg/L) (hs-CRP). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and hs-CRP) are combined to yield a score (0 to no defined upper limit). During Period 2 participants visited study sites at Weeks 28, 32, 36, 40, 44, 48, 52, 56, 60, 64 and 68 or if they discontinued early from the study. A flare was defined as having any 2 consecutive study visits with ASDAS ≥ 2.100.
Time Frame: From Week 28 through 68
Population: Modified Intent-to-treat population: all participants who were randomized into double-blind Period 2 and received at least 1 dose of double-blind study medication; participants with missing data were inputed as nonresponders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 153 | 152
Participants | 72 | 107
Statistical Analysis 1: Comparison: Placebo (Period 2) vs Double-blind Adalimumab (Period 2); Test type: Other; p < 0.001, Chi-squared — 2-sided Pearson's chi-square test

2. Secondary Outcome: Number of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) Inactive Disease at 12 Weeks After Initiation of Rescue Therapy
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of high-sensitivity C-reactive protein (mg/L) (hs-CRP). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and hs-CRP) are combined to yield a score (0 to no defined upper limit). ASDAS Inactive Disease is defined as a score of <1.300.
Time Frame: Rescue Therapy Week 12
Population: Rescued Population: participants with available data who received open-label rescue treatment after the double-blind period
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Period 2): Placebo participants who flared during week 28-68 and received open-label adalimumab 40 mg every other week during the rescue period.
- Double-blind Adalimumab (Period 2): Double-blind adalimumab participants who flared during week 28-68 and received open-label adalimumab 40 mg every other week during the rescue period.
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 37 | 20

3. Secondary Outcome: Number of Participants Achieving ASDAS Major Improvement at 12 Weeks After Initiation of Rescue Therapy
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of high-sensitivity C-reactive protein (mg/L) (hs-CRP). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and hs-CRP) are combined to yield a score (0 to no defined upper limit). ASDAS Major Improvement is defined as a change from baseline ≤ -2.000.
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 21 | 8

4. Secondary Outcome: Number of Participants Achieving ASDAS Clinically Important Improvement at 12 Weeks After Initiation of Rescue Therapy
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of high-sensitivity C-reactive protein (mg/L) (hs-CRP). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and hs-CRP) are combined to yield a score (0 to no defined upper limit). ASDAS Clinically Important Improvement is defined as a change from baseline ≤ -1.100.
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 37 | 17

5. Secondary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 20 Response at 12 Weeks After Initiation of Rescue Therapy
Description: ASAS20 response was defined as improvement of ≥ 20% relative to baseline and absolute improvement of ≥ 1 unit (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 unit) in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 46 | 19

6. Secondary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 40 Response at 12 Weeks After Initiation of Rescue Therapy
Description: ASAS40 response was defined as improvement of ≥ 40% relative to baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 35 | 16

7. Secondary Outcome: Number of Participants Achieving an ASAS 5/6 Response at 12 Weeks After Initiation of Rescue Therapy
Description: An Assessment of Spondyloarthritis International Society (ASAS) 5/6 response is a 20% improvement in 5 out of the following 6 domains:
  * Patient's Global Assessment of disease activity, on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which assesses participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation: the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none) to 10 (very severe/2 hrs or more duration);
  * Spinal mobility: the lateral lumbar flexion score of the Bath AS Metrology Index (BASMI) on a scale from 0 (best mobility) to 10 (worst mobility);
  * High-sensitivity C-reactive protein level (lower levels = less inflammation).
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 63 | 33
Participants | 25 | 9

8. Secondary Outcome: Number of Participants Achieving ASAS Partial Remission at 12 Weeks After Initiation of Rescue Therapy
Description: Assessment in SpondyloArthritis International Society (ASAS) partial remission is defined as an absolute score of < 2 units on a 0 to 10 scale for each of the four following domains:
  * Patient's Global Assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 65 | 36
Participants | 26 | 15

9. Secondary Outcome: Number of Participants Achieving a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at 12 Weeks After Initiation of Rescue Therapy
Description: The Bath Ankylosing Spondylitis (AS) Disease Activity Index assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity. BASDAI50 is a 50% improvement from baseline in BASDAI score.
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Adalimumab (Period 2): Placebo participants who flared during week 28-68 and received open-label adalimumab 40 mg every other week during the rescue period.
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 64 | 34
Participants | 41 | 18

10. Secondary Outcome: Change From Baseline in Disability Index of Health Assessment Questionnaire Modified for the Spondyloarthropathies (HAQ-S) at 12 Weeks After Initiation of Rescue Therapy
Description: Health Assessment Questionnaire modified for spondyloarthropathies (HAQ-S) is a self-reported measure to assess the physical function and health-related quality of life. The Disability Index (DI) of HAQ-S is calculated as the mean of the following 8 category scores (range: 0 [without any difficulty] to 3 [unable to do]): Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Five additional items in the functional status measure were included in the HAQ-S, including carrying heavy packages, sitting for long periods, able to work at a flat topped table, and (if the participant had a driver's license or a car) able to look in the rear view mirror and able to turn head to drive in reverse. The overall score ranges from 0 (no disability) to 3 (very severe, high-dependency disability). Negative mean changes from baseline in the overall score indicate improvement.
Time Frame: Baseline and Rescue Therapy Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 31 | 17
units on a scale | -0.3 (0.55) | -0.4 (0.60)

11. Secondary Outcome: Number of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) Inactive Disease at Weeks 28 and 68
Description: as for outcome 2
Time Frame: Weeks 28 and 68
Population: Period 1 (all enrolled participants who received at least 1 dose of adalimumab); Period 2 (mITT: all randomized participants who received at least 1 dose of double-blind study medication); participants with missing data were inputed as nonresponders.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 323 | 0 | 0
  Week 28 | 295 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 51 | 87

12. Secondary Outcome: Number of Participants Achieving ASDAS Major Improvement at Weeks 28 and 68
Description: as for outcome 3
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 323 | 0 | 0
  Week 28 | 266 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 49 | 89

13. Secondary Outcome: Number of Participants Achieving ASDAS Clinically Important Improvement at Weeks 28 and 68
Description: as for outcome 4
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 323 | 0 | 0
  Week 28 | 316 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 69 | 102

14. Secondary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 20 Response at Weeks 28 and 68
Description: as for outcome 5
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | 315 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 72 | 107

15. Secondary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 40 Response at Weeks 28 and 68
Description: as for outcome 6
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | 302 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 70 | 100

16. Secondary Outcome: Number of Participants Achieving an ASAS 5/6 Response at Weeks 28 and 68
Description: as for outcome 7
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | 253 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 49 | 87

17. Secondary Outcome: Number of Participants Achieving ASAS Partial Remission at Weeks 28 and 68
Description: as for outcome 8
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | 224 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 41 | 64

18. Secondary Outcome: Number of Participants Achieving a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at Weeks 28 and 68
Description: as for outcome 9
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
Participants
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | 317 |  |
  Week 68: number analyzed (Participants) | 0 | 153 | 152
  Week 68 |  | 72 | 103

19. Secondary Outcome: Change From Baseline in Disability Index of Health Assessment Questionnaire Modified for the Spondyloarthropathies (HAQ-S) at Weeks 28 and 68
Description: as for outcome 10
Time Frame: Baseline, Weeks 28 and 68
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label (OL) Adalimumab (Period 1) | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 673 | 153 | 152
units on a scale
  Week 28: number analyzed (Participants) | 324 | 0 | 0
  Week 28 | -0.8 (0.58) |  |
  Week 68: number analyzed (Participants) | 0 | 79 | 112
  Week 68 |  | -0.8 (0.59) | -0.8 (0.63)

20. Secondary Outcome: Time to Flare at Week 68
Description: as for outcome 1
Time Frame: From Week 28 through 68
Population: Modified Intent-to-treat population: all participants who were randomized into double-blind Period 2 and received at least 1 dose of double-blind study medication; participants with missing data were treated as missing.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 153 | 152
weeks | NA [41 to NA] — The survival function was >50%, with an insufficient number of participants with events to estimate median time to flare. The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA. | NA [NA to NA] — The survival function was >50%, with an insufficient number of participants with events to estimate median time to flare. The lower and upper 95% CI limits were not estimable due to an insufficient number of participants with events, indicated by NA.
Statistical Analysis 1: Comparison: Placebo (Period 2) vs Double-blind Adalimumab (Period 2); The statistical test was performed at a 2-sided significance level of 0.05. Time to flare analysis showed statistically significant lower risk of flare in the adalimumab group than in the placebo group; Test type: Other; p < 0.001, Log Rank

21. Secondary Outcome: Time to Partial Flare at Week 68
Description: The Ankylosing Spondylitis Disease Activity Score (ASDAS) tool is a self-administered questionnaire/objective laboratory evaluation. The questionnaire assesses disease activity, back pain, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and duration of morning stiffness on a numeric rating scale (from 0 to 10, with 0 being none and 10 representing a duration of ≥2 hours). The laboratory parameter is a measurement of high-sensitivity C-reactive protein (mg/L) (hs-CRP). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and hs-CRP) are combined to yield a score (0 to no defined upper limit). During Period 2 participants visited study sites at Weeks 28, 32, 36, 40, 44, 48, 52, 56, 60, 64 and 68 or if they discontinued early from the study. A partial flare was defined as having any 2 consecutive study visits with ASDAS ≥ 1.300 but <2.100.
Time Frame: From Week 28 through 68
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 153 | 152
weeks | 41 [41 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA. | 42 [42 to NA] — The upper 95% CI limit was not estimable due to an insufficient number of participants with events, as indicated by NA.

22. Secondary Outcome: Number of Participants Reaching Flare Definition by Week 68
Description: as for outcome 1
Time Frame: From Week 28 through 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 153 | 152
Participants | 81 | 45

23. Secondary Outcome: Number of Participants Reaching Partial Flare Definition by Week 68
Description: as for outcome 21
Time Frame: From Week 28 through 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Period 2) | Double-blind Adalimumab (Period 2)
Number analyzed (Participants) | 153 | 152
Participants | 98 | 62

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 70 days after the last dose of study drug (up to 90 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Open-label (OL) Adalimumab (Period 1), Full Analysis Set: 40 mg every other week (eow), Weeks 0-28. The Full Analysis Set included all participants who enrolled in the open-label period (Period 1) and received at least 1 dose of adalimumab.
- Any Adalimumab Population: The Any Adalimumab Population consisted of all participants who received at least 1 dose of adalimumab any time during the study (including the open-label period, double-blind period and rescue period).
Arm/Group | Open-label (OL) Adalimumab (Period 1), Full Analysis Set | Placebo (Period 2) | Double-blind Adalimumab (Period 2) | Any Adalimumab Population
All-Cause Mortality (participants affected / at risk) | 0/673 | 0/153 | 0/152 | 0/673
Serious Adverse Events (participants affected / at risk) | 19/673 | 10/153 | 1/152 | 28/673
Other Adverse Events (participants affected / at risk) | 221/673 | 51/153 | 57/152 | 275/673
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (OL) Adalimumab (Period 1), Full Analysis Set (N=673) | Placebo (Period 2) (N=153) | Double-blind Adalimumab (Period 2) (N=152) | Any Adalimumab Population (N=673)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
ATYPICAL PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
AXIAL SPONDYLOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
URETHRAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (OL) Adalimumab (Period 1), Full Analysis Set (N=673) | Placebo (Period 2) (N=153) | Double-blind Adalimumab (Period 2) (N=152) | Any Adalimumab Population (N=673)
NASOPHARYNGITIS (Infections and infestations) | 90 (103) | 20 (23) | 25 (32) | 117 (151)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 57 (70) | 12 (14) | 20 (25) | 80 (114)
DIARRHOEA (Gastrointestinal disorders) | 36 (39) | 5 (5) | 6 (7) | 42 (48)
HEADACHE (Nervous system disorders) | 45 (50) | 5 (5) | 7 (7) | 54 (62)
AXIAL SPONDYLOARTHRITIS (Musculoskeletal and connective tissue disorders) | 36 (38) | 21 (23) | 10 (15) | 57 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT01808118/SAP_000.pdf
  • Study Protocol (2015-01-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT01808118/Prot_001.pdf